CLINICAL TRIAL: NCT06883799
Title: Association of Reaction Time and Sleep Quality in Professional Football Players
Status: Completed | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Maciej Kochman, principal investigator, University of Rzeszow
Other Study IDs: 013/04/2024
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Reaction Time; Sport; Football Players; Sleep Quality; Physical Fitness
Keywords: football; reaction time; sleep quality; physical activity; sport; physical fitness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Football players and healthy: The study analyzed 40 football players (study group)
  Interventions: Other: Without intervention.
- healthy, non-trained individuals: healthy, non-trained individuals
  Interventions: Other: Without intervention.

INTERVENTIONS:
Other: Without intervention. — Without intervention

SUMMARY:
Football players need to use their cognitive skills to choose and execute actions in reaction to various stimuli throughout a match and training. Reaction time (RT), an important component of physical fitness, is a key variable for assessing higher cognitive function in football players. For athletes, sleep is also a critical factor influencing sports performance and is widely recognized as a key indicator of overall health. The aim of this study is to assess differences in reaction time and sleep quality as well as the association between these variables in a group of professional football players and a control group. The study analyzes 40 football players (study group) and 40 healthy, non-trained individuals (control group). Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), and reaction times, both simple and complex, are assessed using the AT SMART System reaction speed tester.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, informed written consent to participate in the study
* Minimum of 3 years of experience playing football
* Minimum of 3 training sessions per week
* Age between 18 and 30 years
* No musculoskeletal injuries within the last 6 months
* No disorders or conditions that may affect the study results

Exclusion Criteria:

* Lack of voluntary, informed written consent to participate in the study
* Less than 3 years of experience playing football
* Less than 3 training sessions per week
* Age under 18 or over 30 years
* Presence of musculoskeletal injuries within the last 6 months
* Presence of disorders or conditions that may affect the study results

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Professional football players in the Podkarpackie Voivodeship.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Sleep quality | September 2024
  Pittsburgh sleep quality questionnaire which contained 10 questions about the quality of sleep from the last 4 weeks.
Reaction time | September 2024
  Reaction speed testing was performed using the AT SMART System reaction speed tester. The tester comprises four components: a control panel, a set of manual and foot buttons, a light and sound stimulus indicator, and a power supply.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszów, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No